CLINICAL TRIAL: NCT02242279
Title: Randomised, Double-Blind, Placebo-Controlled, 4-Way Cross-Over Study to Assess the Efficacy and Safety of a Single Dose of Orally Inhaled BEA 2180 BR (Doses 80, 200 and 800 μg) in COPD Patients Followed by an Open-Label, Active-Control (Tiotropium 72 μg)
Brief Title: Study to Evaluate Efficacy and Safety of Inhaled BEA 2180 BR in COPD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1205.3
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

ARMS (5):
- BEA 2180 - low dose (Experimental)
  Interventions: Drug: BEA 2180 BR
- BEA 2180 - medium dose (Experimental)
  Interventions: Drug: BEA 2180 BR; Drug: Placebo
- BEA 2180 - high dose (Experimental)
  Interventions: Drug: BEA 2180 BR
- Tiotropium (Active Comparator)
  Interventions: Drug: Tiotropium
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BEA 2180 BR
  Arms: BEA 2180 - high dose; BEA 2180 - low dose; BEA 2180 - medium dose
Drug: Tiotropium
  Arms: Tiotropium
Drug: Placebo
  Arms: BEA 2180 - medium dose; Placebo

SUMMARY:
Study to investigate the dose-dependent bronchodilator effect and the safety of single inhalation doses of BEA 2180 inhaled via Respimat® compared to placebo in patients with stable Chronic Obstructive Pulmonary Disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

1. All patients have to sign and date an informed consent consistent with International committee on harmonisation (ICH) - Good Clinical Practice (GCP) guidelines prior to participation in the trial, which included medication washout and restrictions
2. All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria:

   Patients must have relatively stable, moderate to severe airway obstruction with an FEV1 ≤ 60% of predicted normal and FEV1 ≤ 70% of FVC (Visits 1 and 2)
3. All patients must have an increase in FEV1 of at least 12% from baseline 45 min after inhalation of 80 μg of ipratropium inhaled via Hydro Fluoro Alkane (HFA) - Metered Dose Inhaler (MDI)
4. Male or female patients 40 years of age or older. Female patients of child bearing potential could not participate in this study
5. Patients must be current or ex-smokers with a smoking history of more than 10 pack/years

   * (Patients who have never smoked cigarettes must be excluded)
6. Patients must be able to perform technically acceptable pulmonary function tests and inhale medication in a competent manner from the Respimat® device and the HandiHaler®

Exclusion Criteria:

1. Patients with significant diseases other than Chronic Obstructive Pulmonary Disease (COPD) must be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
2. Patients with clinically relevant abnormal baseline hematology, blood chemistry, or urinalysis, if the abnormality defines a significant disease
3. Patients with significant prostatic hyperplasia
4. Patients with a recent history (i.e. one year or less) of myocardial infarction
5. Patients with any unstable or life-threatening cardiac arrhythmia or patients who have been hospitalized for such an event within the past year
6. Patients with a history (less than 3 years) of cardiac failure, cor pulmonale or cardiac arrhythmia requiring drug therapy
7. Patients with a malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years. Patients with treated basal cell carcinoma are allowed
8. Patients with known narrow-angle glaucoma
9. Patients with a history of asthma, allergic rhinitis or who have a total blood eosinophil count ≥ 600/mm3. A repeat eosinophil count was not conducted in these patients
10. Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or clinically evident bronchiectasis
11. Patients with known active tuberculosis
12. Patients with a history of and/or active significant alcohol or drug abuse
13. Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons must be excluded
14. Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the Screening Visit (Visit 1)
15. Patients who regularly used daytime oxygen therapy
16. Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to Screening Visit (Visit 1)
17. Patients who are being treated with oral beta-adrenergic
18. Patients who are being treated with beta-blockers
19. Patients who are being treated with cromolyn sodium or nedocromil sodium
20. Patients who are being treated with antihistamines (H1 receptor antagonists), antileukotrienes or leukotriene receptor antagonists for asthma or excluded allergic conditions
21. Patients using oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day
22. Patients with known hypersensitivity to anticholinergic drugs, beta-adrenergic, lactose or any other components of the medication delivery systems
23. Pregnant or nursing women or women of childbearing potential. Female patients have to be either:

    * Surgically sterilized by hysterectomy or bilateral tubal ligation or
    * Post-menopausal for at least two years
24. Patients with previous participation (receipt of randomized treatment) in this study
25. Patients who are participating in another study
26. The randomization of patients with any respiratory infection or COPD exacerbation in the six weeks prior to the Screening Visit (Visit 1) or during the baseline period must be postponed. Patients could be randomized six weeks following recovery from the infection or exacerbation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-06; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Change in Mean Forced Expiratory Volume in 1st second (FEV1) | 23 and 24 hours after single inhalation

SECONDARY OUTCOMES:
Change in FEV1 Area under the concentration-time curve over the respective time interval (AUCtime-interval) | predose, 30, 60 minutes, 2, 3, 4, 6, 8, 10, 12, 23, 24, 26 and 28 hours after inhalation of each single dose
Peak FEV1 | within 3 hours after inhalation of each single dose
Time to peak bronchodilatory response | within 3 hours after inhalation of each single dose
Change in Forced Vital Capacity (FVC) AUCtime-interval | predose, 30, 60 minutes, 2, 3, 4, 6, 8, 10, 12, 23, 24, 26 and 28 hours after inhalation of each single dose
Change in individual FEV1 measurements | up to 71 days
Change in individual FVC measurements | up to 71 days
Number of patients with adverse events | up to 85 days
Area under the plasma concentration-time curve over the respective time interval (AUCtime-interval) | predose, 5 min, 30min, 2 h, 8 h , 24 h
Pre-dose plasma concentration immediately before the inhalation of each single dose (Cpre) | predose
Maximum measured plasma concentration following the inhalation of each single dose (Cmax) | predose, 5 min, 30min, 2 h, 8 h , 24 h
Time from dosing to the maximum plasma concentration the inhalation of each single dose of randomised treatment (tmax) | predose, 5 min, 30min, 2 h, 8 h , 24 h
Amount of unchanged drug excreted over the respective time intervals (Aetime-interval) | predose, 0-4 h, 4-24 h
Renal clearance of the analyte from the time point t1 until the time point t2 (CLR,t1-t2) | predose, 0-4 h, 4-24 h
Fraction of analyte eliminated in urine from different time intervals (fetime-interval) | predose, 0-4 h, 4-24 h
Peak FVC | within 3 hours after inhalation of each single dose